CLINICAL TRIAL: NCT00311298
Title: The Role of Nutritional Support and Diabetes During Treatment of Pulmonary TB: Two Randomized Nutritional Supplementation Trials in Tanzania
Brief Title: Nutrition, Diabetes and Pulmonary TB/HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); The Danish Medical Research Council (Other); Danish Council for Development Research (Other)
Responsible Party: Prof. Henrik Friis, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIMR-UC-2006-01
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Tuberculosis; HIV; Diabetes
Keywords: tuberculosis; hiv; diabetes; protein-energy; micronutrients
MeSH Terms: conditions — Tuberculosis; Diabetes Mellitus; Acquired Immunodeficiency Syndrome | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- No micronutrients (Placebo Comparator): Biscuit without additional micronutrients
  Interventions: Dietary Supplement: Multimicronutrients
- Micronutrients (Experimental): Biscuit with additional micronutrients
  Interventions: Dietary Supplement: Multimicronutrients
- 1 biscuit (Active Comparator): 1 biscuit with micronutrients
  Interventions: Dietary Supplement: Energy and proteins
- 6 biscuits (Experimental): 1 biscuit with micronutrients, plus 5 biscuits without additional micronutrients
  Interventions: Dietary Supplement: Energy and proteins

INTERVENTIONS:
Dietary Supplement: Multimicronutrients — Randomised, double-blind trial among pulmonary TB patients, except those who are found to be sputum positive and HIV positive. Both arms received a daily biscuit weighing 30 g (4.5 g protein, 615 kJ). The biscuit given to the No micronutrient-arm contained no additional micronutrients. The biscuit given to the Micronutrient-arm contained the following micronutrients: vitamin A 5000 IU, vitamin B1 20 mg, vitamin B2 20 mg, vitamin B6 25 mg, vitamin B12 50 microg, folic acid 0.8 mg, niacin 40 mg, vitamin C 200 mg, vitamin E 60 mg, vitamin D3 5 µg / 200 IU, selenium 0.2 mg, copper 5 mg, and zinc 30 mg. The intervention was given for 60 days during initial TB treatment.
  Arms: Micronutrients; No micronutrients
Dietary Supplement: Energy and proteins — Randomised, single-blind trial among sputum-positive HIV-coinfected pulmonary TB patients. Both arms received a daily for biscuit weighing 30 g (4.5 g protein, 615 kJ), with micronutrients (vitamin A 5000 IU, vitamin B1 20 mg, vitamin B2 20 mg, vitamin B6 25 mg, vitamin B12 50 microg, folic acid 0.8 mg, niacin 40 mg, vitamin C 200 mg, vitamin E 60 mg, vitamin D3 5 µg / 200 IU, selenium 0.2 mg, copper 5 mg, and zinc 30 mg). The experimental arm received an additional 5 biscuits without additional micronutrients. Thus, both arms received the same amount of micronutrients. However, the intervention arm received 3690 kJ and 27 g protein per day, while the control arm received 615 kJ and 4.5 g protein. The intervention was given for 60 days during initial TB treatment.
  Arms: 1 biscuit; 6 biscuits

SUMMARY:
We propose a randomised trial among pulmonary TB patients, examined and treated as part of the national TB control programme (WHO, 2003). The aim is to improve TB treatment outcome in high TB and HIV burden countries. The overall objective of the proposed trial is to assess the effect of nutritional support on TB treatment outcomes, and to assess the role of diabetes on risk and severity of TB, and TB treatment outcomes. The study will be conducted in Mwanza Tanzania. All patients will initially be examined for HIV and diabetes. A total of 500 found pulmonary TB smear-positive (PTB+) and HIV positive (HIV+) will be randomised to a daily supplement of 1 versus 6 energy-protein bars throughout treatment, both with full multi-micronutrient (MN) content. A total of 1500 found pulmonary TB smear-negative (PTB-, irrespective of HIV status) and PTB+ and HIV negative (HIV-) will be randomised to 1 daily energy-protein bar containing either low or high MN content.

ELIGIBILITY:
Inclusion Criteria:

* New sputum smear positive or negative pulmonary TB patients

Exclusion Criteria:

* pregnant, terminally ill, other serious diseases (except HIV and diabetes), non-residents

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Weight gain | 2 and 5 months

SECONDARY OUTCOMES:
Grip strength | 2 and 5 months
Arm muscle and arm fat areas | 2 and 5 months
Physical activity | 2 and 5 months
HIV load | 2 months
CD4 count | 2 and 5 months
Serum acute phase reactants | 2 months
Mortality | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Nyagosya Range, MSc, PhD, Principal Investigator — Muhimbili Medical Centre, NIMR; Henrik Friis, MD, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Mwanza Medical Centre, NIMR, Mwanza, Mwanza Region, Tanzania

REFERENCES:
- [Background] Range N, Changalucha J, Krarup H, Magnussen P, Andersen AB, Friis H. The effect of multi-vitamin/mineral supplementation on mortality during treatment of pulmonary tuberculosis: a randomised two-by-two factorial trial in Mwanza, Tanzania. Br J Nutr. 2006 Apr;95(4):762-70. doi: 10.1079/bjn20051684. PMID 16571156
- [Derived] Andersen AB, Range NS, Changalucha J, Praygod G, Kidola J, Faurholt-Jepsen D, Krarup H, Grewal HM, Friis H. CD4 lymphocyte dynamics in Tanzanian pulmonary tuberculosis patients with and without HIV co-infection. BMC Infect Dis. 2012 Mar 21;12:66. doi: 10.1186/1471-2334-12-66. PMID 22436147
- See also: National Institute of Medical Research — http://www.nimr.or.tz/